CLINICAL TRIAL: NCT03517891
Title: Intervention to Promote Physical Activation and Improve Sleep and Feeding Practices in Infants for Preventing Obesity Early in Life (The Baby-Act Trial)
Brief Title: The Baby Act Trial (BAT): a Multimodal Lifestyle Intervention
Acronym: BAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Puerto Rico (Other)
Collaborators: Marshfield Clinic Research Foundation (Other); Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A4540117
Record Dates: First submitted 2018-04-20; First posted 2018-05-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-05

CONDITIONS: Obesity in Childhood
Keywords: Physical activity; Sleep pattern; Nutrition; Education
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial in 16 WIC clinics. We will randomly assign 8 clinics to the intervention arm and 8 to control (usual care) arm. The intervention will combine key messages and activities designed to promote sound parenting skills that support and sustain healthy lifestyles beginning at birth until the infant is 12 months of age. Participants will be recruited at the WIC clinics during in the last trimester of pregnancy. The primary, intention-to-treat, analysis will evaluate the effect of the intervention on excessive weight gain and rate of weight gain from birth until 12 months. The intention-to-treat approach will allow us to evaluate the expected effect of adding the proposed intervention to the current WIC curriculum. Secondary analyses will include effects of the intervention on objective measures of infant activation, sedentary behaviors and sleep, diet quality, and feeding practices.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: We will use a random allocation process for each clinic with the exception of the 2 satellite clinics which will be randomly assigned separately to ensure assignment of 1 satellite clinic per treatment arm. Additional attention to the distribution of the satellite clinics is deemed necessary as the flow of participants at these sites differs from other clinics due to extended working hours and location of facilities (shopping malls). Randomization will take into account the number of pregnant participants per clinic as well as breastfeeding statistics as an important determinant of future infant obesity. Changes in clinic location and service hours have been documented during the course of the study to account for operational changes implemented by our community partner in response to extraordinary events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WIC + (Experimental): The intervention consist in the implementation of an enhanced nutritional education and services model through the use of a combination of modalities to disseminate messages and educational materials framed in the health empowerment model. Each component of the intervention has been developed to provide the information consistent with the theoretical framework of the modality being used.
  The intervention targets the following behaviors: Infant activation, Healthy sleep patterns, Screen time, Healthy feeding practices.
  Interventions: Behavioral: WIC+
- WIC Standard of care (Control) (No Intervention): Participants recruited in randomly assigned control clinics will receive the WIC program standard of care. This includes the projected implementation of a web page for the nutritional education contacts. We will update our definition of the PR WIC program standard of care upon recruitment initiation and throughout the study implementation phase. We will also document the utilization rate of the web base platform provided by WIC among the control participants to determine baseline use of distance learning platforms.

INTERVENTIONS:
Behavioral: WIC+ — intervention was based on the Health Self-Empowerment Theory. It will be adapted for the web-based platform using the Persuasive Technology and Persuasive System Design models. These models focus on the human-computer interface and how technology can/is used as a persuasive tool for behavior change. We will also include Bandura's Social Cognitive Theory.
  The intervention will be delivered through the combination of:
  educational modules provided through an interactive distance learning platform designed to provide learning experiences using multiple modalities; short messaging platforms to promote adoption of healthy behaviors and use of the educational platform; one to one sessions with the interventionist over the telephone.
  Arms: WIC +

SUMMARY:
Childhood obesity is increasing, particularly among Hispanics. Rapid weight gain during childhood increases the risk of obesity in childhood and in adulthood, also increasing the risk of chronic diseases such as diabetes and hypertension. This can be prevented with interventions during early in life that address multiple risk factors associated with the early development of obesity. Therefore, the purpose of this study is to test an intervention to promote baby activation and improve their sleep patterns and feeding patterns from birth to 12 months of age. For this purpose, pregnant women participating in the Special Nutrition Women, Infants and Children (WIC) Program in Puerto Rico will be recruited and randomly assigned to the control group (usual care within the program) or to the WIC + group (usual care + intervention). The intervention will focus on age-appropriate physical activity for children, healthy sleep and limited time on the screen, healthy dietary patterns and growth monitoring. The content will be delivered with a multimedia approach (web platform, mobile messages and telephone follow-up). If successful, this intervention could be adopted by the WIC program in Puerto Rico to help prevent childhood obesity among its participants. This will help improve the health of minorities and eliminate health disparities among Hispanics and other at-risk groups.

DETAILED DESCRIPTION:
Infant obesity is increasing in the US, particularly among Hispanics. Rapid weight gain during critical periods of infancy increases the risk of obesity in childhood, continuing into adulthood. This could be prevented through multifaceted programs that address multiple risk factors (e.g., physical activity, sleep, eating behaviors and parental skills). Evidence on successful lifestyle interventions for childhood obesity prevention often promote a comprehensive approach delivered at multiple levels (i.e., individual, family, and community) and delivered through population-level programs. One such program is The Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). WIC serves low-income women who are pregnant and/or have infants and/or young children, groups that are among those at the greatest risk of early weight gain. Our long-term goal is to prevent infant obesity through a structured curriculum that provides a combination of key messages and activities designed to promote sound parenting skills that support and sustain healthy lifestyle (i.e., developmentally appropriate exercises for 'infant activation', sleep and healthy eating behavior) beginning at birth. The proposed intervention is an integrated novel approach leveraging current WIC outreach practices and technology for complementing the current standard of care of the WIC Program. The investigators will assess the clinical effectiveness of this novel complementary intervention among caregivers of infants (0 and 12 months) who are participants of the Puerto Rico WIC program through a cluster-randomized controlled trial in 20 WIC clinics located within the San Juan Metropolitan Area of Puerto Rico. In this design, an equal number of clinics will be randomized to the control or intervention arm. The lifestyle intervention will focus on age-appropriate infant's physical activation, healthy sleep and sedentary patterns, and healthy diet quality, by improving parenting skills. Intervention content will be delivered through a combination of technology (multi-media computer-based platforms and mobile messages) and individual counseling (phone and in-person follow-up). Participation in the intervention will begin during the last trimester of pregnancy and will continue until the infant is 12 months of age. The investigators have already tested the information of such an intervention among a small group of 10 mother-infant dyads during their first year of life, with excellent acceptability. Our main outcome is infant rate of weight gain at 12 months of age. Secondary outcomes include: 1) lifestyle behaviors, such as objectively measured hours of infant movement, sedentary behaviors and sleep; 2) diet quality score (which includes breastfeeding and amount of intake of each food group); 3) other feeding practices (i.e. spoon-feeding, addition of foods to the bottle). The research plan also includes a detailed evaluation of the cost of the intervention as a modification of the current WIC curriculum.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit pregnant women age 18 years and older who are participants of the WIC program that:

  1. are in the 3rd trimester,
  2. intend to enroll their infant in the WIC program when he/she is born,
  3. are experiencing singleton pregnancies;
  4. agree to participate independently of the assigned group; and 5) can read and have access to the internet.

Exclusion Criteria:

* We will exclude pregnant women that:

  1. report high risk pregnancies (history of hypertension of any type, diabetes of any type, antenatal diagnosis of intrauterine growth failure or major congenital anomalies);
  2. who plan to leave their WIC clinic within the study time frame; and
  3. a history of emotional or mental health disorders that would preclude active participation in the study. Also newborns who are premature (before week 37 of gestation), with developmental disabilities, with severe conditions such as hypoxic ischemic encephalopathy, feeding disorders, intractable seizures or any other severe neurologic or muscular disorders and metabolic diseases that require specialized diet, and those requiring prolonged hospitalization at birth (>7 days) will also be excluded from participation once the diagnosis is achieved.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Adequate weight gain during first year | one year
  The main study outcome is adequate weight gain based on gender adjusted Z score using the World Health Organization weight (kilogram) for length (centimeter) growth curves.

SECONDARY OUTCOMES:
Objective assessment of infant activity. | 0-1 month, 6 months, 1 year
  Infant movement and activity patterns will be evaluated using accelerometry data.
Objective sleep measures | 0-1 month, 6 months, 1 year
  Accelerometry data will be analyzed to assess sleep patterns in infants.
General Infant Feeding Practices Questionnaire | 0-1 month, 6 months, 1 year
  This will be assessed from the General Feeding Practices Questionnaire completed at each assessment visit. This instrument was developed to document breastfeeding practices, time of introduction of foods and the presence of other stimuli while feeding.
Diet quality | 0-1 month, 6 months, 1 year
  This will be measured using a validated infant Food Frequency Questionnaire, which will be completed at each assessment visit. The infant food frequency questionnaire was developed to document the food provided to infants 0 to 24 months of age. Information collected allows for calorie and nutrient content assessment and comparison to established nutritional guidelines.
Rate of infant growth. | Birth, 1 month, 6 months, 1 year
  Difference in gender and age adjusted weight for length Z scores determined using the World Health Organization growth curves at each assessment time-point will be evaluated to determine the impact of the intervention.
Reported measures of physical activity | 0-1 month, 6 months, 1 year
  Participants will be asked to complete a survey to document the activities and the time spent performing the activities taught as part of the intervention.
Reported measures of sleep | 0-1, 6 months, 1 year
  Participants will be asked to complete a survey to document characteristics of their infant's sleep pattern and duration of sleep periods.
Weight | 0-1 months, 6 months, 1 year
  The infant's weight will be documented in kilograms at every study assessment time-point and evaluated using the World Health Organization gender appropriate growth curves.
Length | 0-1 months, 6 months, 1 year
  The infant's Length will be documented in centimeters at every study assessment time-point and evaluated using the World Health Organization gender appropriate growth curves.
Head Circumference | 0-1 months, 6 months, 1 year
  As part of the growth assessment the infant's head circumference will be documented in centimeters at every study assessment time-points.
Social determinants of health. | 1 year
  We have added constructs of social capital to our exit interview and integrated the Accountable Health Communities Health-Related Social Needs 10-item screening tool.
Infant Oral Health | 1 year
  We are collecting self reported data related to oral health care and dentition among infants.

OTHER OUTCOMES:
Per participant cost of providing the intervention | 1 year
  Aggregate cost of the implementation of the intervention will be determined including the direct costs of maintaining the distance learning and messaging platforms as well as the personnel cost.
Dried blood spot sample collection | 0-1 and 12 Months
  Participants will be offered the opportunity to donate a sample of capillary blood collected in dried blood spots. Samples will be stored for future analysis including but not limited to metabolic (nutritional biomarkers including vitamins and lipid profiles), inflammatory, oxidative stress biomarkers as well as contribute to epigenetic assessments of lifestyle intervention trials of this currently understudied and genetically admixed population.
Saliva and stool samples | 0-1, 3, 6 and 12 months
  Participants will be offered the opportunity to donate samples from their infants for microbiome and metabolome assessment in future studies. This is an optional study procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Maribel Campos, MD MSc MBA, Principal Investigator — University of Puerto Rico Medical Sciences Campus; Cristina Palacios, PhD MS, Principal Investigator — Florida International University; Jeremy Pomeroy, PhD, Principal Investigator — Marshfield Clinic Research Institute
Locations (1):
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will gather data on the effects of a lifestyle intervention to prevent infant obesity: self-reported socio-demographics, lifestyles, health-related variables, compliance to the intervention, anthropometrics. Results have been presented to the Center for Collaborative Health Disparities Research (CCRHD) and National Institute of Minority Health and Health Disparities (NIMHD) Officials regularly. Findings will be reported at Program Project Meetings and other scientific meetings and published in peer-reviewed journals. Data will not be disseminated outside the University of Puerto Rico until the established study outcome measures have been published. Summary data statistics, publication analysis and any other supplementary data will be posted on the Center for Collaborative Health Disparities Research.
Supporting Information: Study Protocol, SAP
Time Frame: De identified data sets and supporting documents will be made available to the scientific community once established outcomes measures have been published.
Access Criteria: Research proposal must be approved by the PIs and the University of Puerto Rico Medical Sciences Campus Institutional Review Board (UPR-MSC IRB). We will only provide access to de-identified data required to address the proposed research goals. We will make the data, repository samples and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Criteria are subject to review. PIs will publish any additional requirements or criteria associated to the management of data request as emerging regulations or resource limitations might require revision of this plan.

REFERENCES:
- [Background] Campos M, Pomeroy J, Mays MH, Lopez A, Palacios C. Intervention to promote physical activation and improve sleep and response feeding in infants for preventing obesity early in life, the baby-act trial: Rationale and design. Contemp Clin Trials. 2020 Dec;99:106185. doi: 10.1016/j.cct.2020.106185. Epub 2020 Oct 22. PMID 33099015
- [Derived] Kallis Colon MG, Lopez A, Campos Rivera M, Pomeroy J, Palacios C. Baby-Act Intervention to Prevent Excessive Infant Weight Gain: Development, Implementation, Lessons Learned, and Future Applications. Matern Child Health J. 2025 Apr;29(4):572-581. doi: 10.1007/s10995-025-04082-x. Epub 2025 Mar 22. PMID 40120064